CLINICAL TRIAL: NCT07042971
Title: A Multicenter, Randomized Controlled Trial of Pre-operative BiPAP Training and Post-extubation BiPAP Support to Reduce Peri-operative Tracheostomy or Re-intubation in Patients at High Risk for Bilateral Vocal-Cord Paralysis
Brief Title: Peri-operative BiPAP to Prevent Tracheostomy in High-Risk Bilateral Vocal-Cord Paralysis (BVCP)
Acronym: BVCP-BiPAP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, Director & Head of Thyroid Surgery, Principal Investigator, Clinical Professor, Fujian Medical University Union Hospital
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Diagnostic
Other Study IDs: BVCP-BiPAP
Record Dates: First submitted 2025-06-21; First posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Vocal Cord Paralysis, Bilateral; Airway Obstruction, Postoperative; Thyroid Neoplasms; Sleep Apnea, Obstructive
Keywords: BiPAP; Non-invasive Ventilation; Continuous Positive Airway Pressure; Peri-operative Airway Management; Tracheostomy Avoidance; Thyroidectomy; Neck Surgery; Glottic Stenosis; Pre-operative Sleep Training; Voice Handicap Index
MeSH Terms: conditions — Vocal Cord Paralysis; Airway Obstruction; Thyroid Neoplasms; Sleep Apnea, Obstructive

STUDY DESIGN:
Intervention Model Description: Two-by-two factorial randomized controlled trial testing the independent and combined effects of (A) 7-day pre-operative BiPAP training and (B) immediate post-extubation BiPAP support.
Masking Description: Open-label; blinding not feasible because BiPAP mask/pressures are apparent. Primary endpoint (tracheostomy or re-intubation) is objective.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (4):
- Training + Post-op BiPAP (Experimental): Participants receive 7-day Pre-operative BiPAP Training and Post-extubation BiPAP Support for ≥ 48 h after surgery.
  Interventions: Device: Post-extubation BiPAP Support; Other: Standard Peri-operative Care
- Training Only (Experimental): Participants receive 7-day Pre-operative BiPAP Training. No routine BiPAP after extubation; peri-operative care otherwise standard.
  Interventions: Other: Standard Peri-operative Care
- Post-op BiPAP Only (Experimental): No pre-op training. BiPAP started immediately after extubation and continued ≥ 48 h.
  Interventions: Device: Pre-operative BiPAP Training; Device: Post-extubation BiPAP Support
- Standard Care (Active Comparator): No planned BiPAP. Airway managed with institutional standard care only.
  Interventions: Device: Pre-operative BiPAP Training; Other: Standard Peri-operative Care

INTERVENTIONS:
Device: Pre-operative BiPAP Training — Seven consecutive nights (≥ 4 h/night) of BiPAP use at home or on ward, pressure ladder EPAP 6→8 cmH₂O / IPAP 12→16 cmH₂O, recorded on SD card; devices: ResMed AirCurve 10 ST or Philips A40.
  Arms: Post-op BiPAP Only; Standard Care
Device: Post-extubation BiPAP Support — Same BiPAP device started immediately after tracheal extubation; EPAP 8 cmH₂O / IPAP 14 cmH₂O (or patient's final training setting) maintained ≥ 48 h, then weaned when SpO₂ ≥ 94 % off-BiPAP for 24 h.
  Arms: Post-op BiPAP Only; Training + Post-op BiPAP
Other: Standard Peri-operative Care — Routine oxygen, nebulized steroids, airway monitoring; rescue re-intubation or tracheostomy per institutional protocol; no planned BiPAP unless crossover criteria met.
  Arms: Standard Care; Training + Post-op BiPAP; Training Only

SUMMARY:
Why: After thyroid or neck surgery, some patients can lose movement of both vocal cords (bilateral vocal-cord paralysis, BVCP). This can make breathing difficult and often leads to an emergency or preventive tracheostomy ("wind-pipe") surgery.

What: This study will test two simple ways to avoid a tracheostomy:

Pre-operative BiPAP sleep training - patients practice sleeping with a non-invasive BiPAP breathing machine for seven nights before surgery so they become comfortable with the mask and pressures.

Immediate post-extubation BiPAP support - the same BiPAP machine is started as soon as the breathing tube is removed in the operating room or recovery area.

How: Adults (18-80 years) who already have, or are at high risk of getting, BVCP will be randomly assigned to one of four groups in a 2 × 2 design:

• Group 1: training + post-op BiPAP • Group 2: training only • Group 3: post-op BiPAP only • Group 4: standard care (no planned BiPAP).

Main goal: To find out whether either or both BiPAP strategies reduce the need for tracheostomy or re-intubation during the first 7 days after surgery.

What participants do: Eligible patients will undergo routine surgery plus the assigned BiPAP plan. Breathing events, comfort, hospital stay, and voice quality will be recorded up to 6 months.

Potential benefit/risk: BiPAP is non-invasive and already FDA-cleared for home and hospital use, but some people may feel mask discomfort or air leaks. Trained staff will adjust settings and stop BiPAP if serious problems occur.

DETAILED DESCRIPTION:
Background and Rationale Bilateral vocal-cord paralysis (BVCP) after thyroid and neck procedures poses an immediate risk of airway obstruction. Historical management favors prophylactic or rescue tracheostomy; however, tracheostomy carries morbidity, cost, and long-term stigma. Case series suggest that non-invasive ventilation (NIV) using BiPAP can stent the glottic opening while providing ventilatory support, but no prospective randomized data exist.

Objectives Primary: Compare the 7-day composite rate of (a) tracheostomy or (b) re-intubation among patients managed with (i) pre-operative BiPAP training, (ii) immediate post-extubation BiPAP, both, or neither.

Secondary: BiPAP usage hours, hypoxemic events, ICU/hospital length of stay, Voice Handicap Index-10 (VHI-10) and Eating Assessment Tool-10 (EAT-10) scores, normalized glottic area (NGA %) at 6 months, cost.

Study Design Multicenter, open-label, factorial (2 × 2) randomized controlled trial. Randomization (block size = 4) stratified by center. Total planned enrollment: 204 (to allow for 10 % attrition), yielding ~46 evaluable participants per arm.

Interventions Pre-operative BiPAP training: nightly ≥ 4 h for 7 consecutive nights, pressure ladder EPAP 6 → 8 cmH₂O / IPAP 12 → 16 cmH₂O, recorded on SD-card.

Post-extubation BiPAP: same machine and pressures applied immediately after extubation and continued ≥ 48 h or until patient maintains SpO₂ ≥ 94 % for 24 h without BiPAP.

Standard care includes oxygen, nebulization, steroids, and surgical airway if necessary.

Eligibility (key points) Inclusion: age 18-80; scheduled thyroid/neck surgery; pre-op fixed cords at midline/paramedian or glottic gap ≤ 3 mm OR ≥ 2 high-risk factors (bilateral neck re-entry, tumor near both RLNs, bilateral C + L lymph-node dissection, severe OSA AHI ≥ 30, BMI ≥ 30).

Exclusion: emergency surgery, existing tracheostomy, ventilator dependence, mask intolerance, pregnancy, inability to consent.

Outcomes and Assessments

* Airway status monitored continuously POD 0-2, then daily to POD 7.
* ABG, pulse oximetry, and flexible laryngoscopy performed per protocol schedule.
* Adverse events graded by CTCAE v5.0; DSMB halting rule: ≥ 3 grade 3 airway failures in any arm.

Statistical Methods Intention-to-treat for primary endpoint. Log-binomial regression with center as random effect to estimate risk ratios for each main effect and their interaction. Kaplan-Meier curves for "tracheostomy-free survival." Interim analysis at 50 % information using O'Brien-Fleming alpha-spending.

Regulatory Status Devices (ResMed AirCurve 10 ST; Philips A40) are FDA-cleared class II ventilators (510(k)); IRB classified study as non-significant-risk device research exempt from IDE under 21 CFR 812.2(b).

Data Sharing De-identified individual participant data and statistical code will be shared upon reasonable request 6 months after final publication.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 - 80 years.
* Scheduled for thyroidectomy or other neck surgery under general anesthesia.
* High risk of bilateral vocal-cord paralysis (BVCP) defined by at least ONE of:

  * Pre-operative flexible laryngoscopy showing fixed vocal cords at midline or paramedian position, or glottic gap ≤ 3 mm; OR
  * Presence of ≥ 2 high-risk factors:

    * Planned bilateral central plus lateral neck dissection
    * Re-operative bilateral neck surgery or dense scarring
    * Tumor involving both recurrent laryngeal nerves or crico-arytenoid joints
    * Severe obstructive sleep apnea (AHI ≥ 30 events/hour)
    * Body-mass index (BMI) ≥ 30 kg/m²
* Able to tolerate and give informed consent for BiPAP mask use.

Exclusion Criteria:

* Emergency surgery or need for immediate tracheostomy.
* Existing tracheostomy or home ventilator dependence.
* Inability to protect airway (e.g., Glasgow Coma Scale < 13).
* Craniofacial anomaly or skin condition precluding mask seal.
* Pregnancy or breastfeeding.
* Participation in another interventional trial that could interfere with study endpoints.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Composite "Airway Failure" (Tracheostomy OR Re-intubation) | The first occurrence of (a) surgical tracheostomy or (b) endotracheal re-intubation for respiratory distress within 7 days after extubation. Event status adjudicated by an independent investigator using pre-defined criteria.
  Post-operative Day 0 through Day 7

SECONDARY OUTCOMES:
Total BiPAP Usage Hours | Post-op Day 0 to Day 2 (48 hours)
  Sum of hours recorded by device SD-card while patient is connected to BiPAP during the first 48 h after extubation.
Hypoxemic Episodes (SpO₂ < 90 % ≥ 3 min) | Post-op Day 0 to Day 2
  Number of discrete desaturation events captured by continuous pulse oximetry logs.
ICU Length of Stay | Surgery end → ICU discharge (up to 7 days)
  Hours from ICU admission to ICU discharge documented in EMR.
Voice Handicap Index-10 (VHI-10) | 6 months (±14 days) post-op
  Patient-reported outcome; total score 0-40 (higher = worse voice handicap).
Normalized Glottic Area (NGA %) | Baseline pre-op and 6 months post-op
  Percentage of glottic opening area measured on flexible laryngoscopy and normalized to true-vocal-fold length.

CONTACTS AND LOCATIONS:
Overall Officials: Bo WANG, MD, Principal Investigator — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, FJ, China

IPD SHARING:
Plan to Share IPD: Undecided